CLINICAL TRIAL: NCT01993329
Title: A Randomised, Double-Blind, Double-Dummy, Placebo-Controlled, Three-Way Cross-over Study to Evaluate the Effect of AF-219 on Methacholine Hyper-Reactivity in Subjects With Asthma
Brief Title: A Study to Evaluate the Effect of Gefapixant (AF-219/MK-7264) on Methacholine Hyper-reactivity in Participants With Asthma (MK-7264-009)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Afferent Pharmaceuticals, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7264-009; AF219-009 (Other: Afferent Pharmaceuticals); 2013-003566-13 (EudraCT Number); MK-7264-009 (Other: Merck)
Record Dates: First submitted 2013-11-15; First posted 2013-11-25 (Estimated); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Gefapixant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Gefapixant 50/ Gefapixant 300/ Placebo (Experimental): Gefapixant 50 mg and placebo (for gefapixant 300 mg) twice daily for 3.5 days during Period 1, gefapixant 300 mg and placebo (for gefapixant 50 mg) twice daily for 3.5 days during Period 2, placebo to match gefapixant 50 mg and placebo to match gefapixant 300 mg twice daily for 3.5 days during Period 3. Each period is separated by at least a 7-day wash-out period.
  Interventions: Drug: Gefapixant 50 mg; Drug: Gefapixant 300 mg; Drug: Placebo to mimic 50 mg tablets; Drug: Placebo to mimic 300 mg tablets
- Gefapixant 50/ Placebo/ Gefapixant 300 (Experimental): Gefapixant 50 mg and placebo (for gefapixant 300 mg) twice daily for 3.5 days during Period 1, placebo to match gefapixant 50 mg and placebo to match gefapixant 300 mg twice daily for 3.5 days during Period 2, gefapixant 300 mg and placebo (for gefapixant 50 mg) twice daily for 3.5 days during Period 3. Each period is separated by at least a 7-day wash-out period.
  Interventions: Drug: Gefapixant 50 mg; Drug: Gefapixant 300 mg; Drug: Placebo to mimic 50 mg tablets; Drug: Placebo to mimic 300 mg tablets
- Gefapixant 300/ Gefapixant 50/ Placebo (Experimental): Gefapixant 300 mg and placebo (for gefapixant 50 mg) twice daily for 3.5 days during Period 1, gefapixant 50 mg and placebo (for gefapixant 300 mg) twice daily for 3.5 days during Period 2, placebo to match gefapixant 50 mg and placebo to match gefapixant 300 mg twice daily for 3.5 days during Period 3. Each period is separated by at least a 7-day wash-out period.
  Interventions: Drug: Gefapixant 50 mg; Drug: Gefapixant 300 mg; Drug: Placebo to mimic 50 mg tablets; Drug: Placebo to mimic 300 mg tablets
- Gefapixant 300/ Placebo/ Gefapixant 50 (Experimental): Gefapixant 300 mg and placebo (for gefapixant 50 mg) twice daily for 3.5 days during Period 1, placebo to match gefapixant 50 mg and placebo to match gefapixant 300 mg twice daily for 3.5 days during Period 2, gefapixant 50 mg and placebo (for gefapixant 300 mg) twice daily for 3.5 days during Period 3. Each period is separated by at least a 7-day wash-out period.
  Interventions: Drug: Gefapixant 50 mg; Drug: Gefapixant 300 mg; Drug: Placebo to mimic 50 mg tablets; Drug: Placebo to mimic 300 mg tablets
- Placebo/ Gefapixant 50/ Gefapixant 300 (Experimental): Placebo to match gefapixant 50 mg and placebo to match gefapixant 300 mg twice daily for 3.5 days during Period 1, gefapixant 50 mg and placebo (for gefapixant 300 mg) twice daily for 3.5 days during Period 2, gefapixant 300 mg and placebo (for gefapixant 50 mg) twice daily for 3.5 days during Period 3. Each period is separated by at least a 7-day wash-out period.
  Interventions: Drug: Gefapixant 50 mg; Drug: Gefapixant 300 mg; Drug: Placebo to mimic 50 mg tablets; Drug: Placebo to mimic 300 mg tablets
- Placebo/ Gefapixant 300/ Gefapixant 50 (Experimental): Placebo to match gefapixant 50 mg and placebo to match gefapixant 300 mg twice daily for 3.5 days during Period 1, gefapixant 300 mg and placebo (for gefapixant 50 mg) twice daily for 3.5 days during Period 2, gefapixant 50 mg and placebo (for gefapixant 300 mg) twice daily for 3.5 days during Period 3. Each period is separated by at least a 7-day wash-out period.
  Interventions: Drug: Gefapixant 50 mg; Drug: Gefapixant 300 mg; Drug: Placebo to mimic 50 mg tablets; Drug: Placebo to mimic 300 mg tablets

INTERVENTIONS:
Drug: Gefapixant 50 mg — Gefapixant 50 mg tablet administered orally
  Other Names: AF-219; MK-7264
Drug: Gefapixant 300 mg — Gefapixant 300 mg tablet administered orally
  Other Names: AF-219; MK-7264
Drug: Placebo to mimic 50 mg tablets — Sugar pill manufactured to mimic gefapixant 50 mg tablets
Drug: Placebo to mimic 300 mg tablets — Sugar pill manufactured to mimic gefapixant 300 mg tablets

SUMMARY:
This is a randomized, double-blind, double-dummy, placebo-controlled, three-way cross-over, single centre study in participants with asthma undergoing inhalation of methacholine and adenosine triphosphate (ATP) to assess the provocative concentration (PC20) response of two dose levels of gefapixant (AF-219) compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Women of child-bearing potential (WOCBP) (i.e., women who are not surgically sterile, not having had hysterectomy, bilateral tubal occlusion or bilateral oophorectomy, or are not postmenopausal) must have a negative pregnancy test at Screening and prior to randomization. WOCBP must be using 2 forms of acceptable birth control method from Screening through the Follow-Up Visit. Acceptable birth control methods include (of which 2 must be used):

  * Established use of oral, injected or implanted hormonal methods of contraception
  * Intrauterine device (IUD) or intrauterine system (IUS)
  * Condom with spermicide
  * Diaphragm with spermicide
  * Double-barrier method (diaphragm for female participant and condom for male partner with spermicidal) satisfies the requirement for 2 forms of acceptable birth control. When in line with the preferred lifestyle of the participant, true and complete abstinence (not periodic abstinence) is acceptable.
  * Male participants with partners WOCBP (as defined in Inclusion No. 2) must use 2 methods of acceptable birth control with their partner, 1 of which must be a barrier method. Contraception must start from screening and continue until 3 months after last dose of study drug.
* Non-smokers or former smokers, who stopped smoking 6 months prior to screening. Former smokers should not have a smoking history of more than 5 pack years (1 pack of 20 cigarettes per day over 5 years).
* Physician documented history or diagnosis of asthma for at least 6 months prior to screening according to the Global Initiative in Asthma guidelines (GINA, 2012).
* Requires the use of Short acting β2-agonist therapy only (≤ 8 puffs per day) for at least 4 weeks prior to screening and prior to randomization.

Exclusion Criteria:

* Has been hospitalized or attended the emergency department for an asthma attack in the 12 months prior to screening.
* Exacerbation of asthma or lower respiratory tract infection during the 4 weeks before screening or prior to randomization.
* Upper respiratory tract infection during the 4 weeks before screening or prior to randomization requiring treatment with antibiotics.
* Inhaled or systemic corticosteroids (oral, intravenous, intramuscular) within 4 weeks prior to screening or prior to randomization.
* Short-acting or long-acting antihistamines within 48hrs or 7 days, respectively, prior to screening.
* Body mass index (BMI) <18 kg/m2 or ≥ 35 kg/m2 at screening.
* History of kidney/bladder stones (nephro/uro-lithiasis) within 5 years of screening.
* History of conditions or disorders that predispose to nephrolithiasis, such as Type 1 renal tubular acidosis, cystinuria, gout, hyperparathyroidism, inflammatory bowel disease (i.e., ulcerative colitis and Crohn's disease), short bowel syndrome, or bariatric surgery.
* History of concurrent malignancy or recurrence of malignancy within 2 years prior to Screening (not including participants with basal cell carcinomas or cervical carcinoma in situ that has been successfully treated surgically).
* Personal or family history of congenital long QT Interval on ECG (QT) syndrome.
* Presence of a cardiac pacemaker.
* History of a diagnosis of drug or alcohol dependency or abuse within approximately the last 3 years.
* Diagnosis of depression, psychosis, bipolar disorder, or schizoaffective disorder.
* Participants with diabetes Type I or uncontrolled diabetes Type II or Glycosylated Hemoglobin (HbA1c) > 8.0% at screening.
* Any condition possibly affecting drug absorption e.g., gastrectomy, gastroplasty, any type of bariatric surgery, vagotomy, or bowel resection.
* History of cutaneous adverse drug reaction to sulphonamides or signs or symptoms suggestive of anaphylaxis to sulphonamides.
* Requiring concomitant therapy with prohibited medications at screening or prior to randomization.
* Pregnant or breastfeeding woman.
* Donation of sperm from Screening until 3 months after the last dose of study drug.
* Male participants with pregnant female partners.
* Treatment with an investigational drug within 30 days or five half-lives preceding the first dose of study medication or plans to take another investigational drug within 30 days of study completion.
* Donation or loss of 400 mL or more of blood or donations of plasma within eight (8) weeks prior to initial dosing or longer if required by local regulation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2014-02-20 (Actual); Study Completion 2014-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Afferent Pharmaceuticals, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A Screening Phase of up to 21 days ensured that each participant met all the specified inclusion and none of the exclusion criteria. Screening procedures were performed over at least 2 days
Groups:
- Gefapixant 50 mg>Gefapixant 300 mg>Placebo: Gefapixant 50 mg twice daily (BID) on Days 1-3 and once daily in the morning Day 4 in Period 1, followed by a washout period of ≥7 days, then Gefapixant 300 mg BID on Days 1-3 and once daily in the morning Day 4 in Period 2 followed by a washout period of ≥7 days, then Placebo BID on Days 1-3 and once daily in the morning Day 4 in Period 3
- Gefapixant 50 mg>Placebo>Gefapixant 300 mg: Gefapixant 50 mg BID on Days 1-3 and once daily in the morning Day 4 in Period 1, followed by a washout period of ≥7 days, then Placebo BID on Days 1-3 and once daily in the morning Day 4 in Period 2, followed by a washout period of ≥7 days, then Gefapixant 300 mg BID on Days 1-3 and once daily in the morning Day 4 in Period 3
- Gefapixant 300 mg>Gefapixant 50 mg>Placebo: Gefapixant 300 mg BID on Days 1-3 and once daily in the morning Day 4 in Period 1, followed by a washout period of ≥7 days, then Gefapixant 50 mg BID on Days 1-3 and once daily in the morning Day 4 in Period 2, followed by a washout period of ≥7 days, then Placebo BID on Days 1-3 and once daily in the morning Day 4 in Period 3
- Gefapixant 300 mg>Placebo>Gefapixant 50 mg: Gefapixant 300 mg BID on Days 1-3 and once daily in the morning Day 4 in Period 1, followed by a washout period of ≥7 days, then Placebo BID on Days 1-3 and once daily in the morning Day 4 in Period 2, followed by a washout period of ≥7 days, then Gefapixant 50 mg BID on Days 1-3 and once daily in the morning Day 4 in Period 3
- Placebo> Gefapixant 50 mg>Gefapixant 300 mg: Placebo BID on Days 1-3 and once daily in the morning Day 4 in Period 1, followed by a washout period of ≥7 days, then Gefapixant 50 mg BID on Days 1-3 and once daily in the morning Day 4 in Period 2, followed by a washout period of ≥7 days, then Gefapixant 300 mg BID on Days 1-3 and once daily in the morning Day 4 in Period 3
- Placebo> Gefapixant 300 mg>Gefapixant 50 mg: Placebo BID on Days 1-3 and once daily in the morning Day 4 in Period 1, followed by a washout period of ≥7 days, then Gefapixant 300 mg BID on Days 1-3 and once daily in the morning Day 4 in Period 2, followed by a washout period of ≥7 days, then Gefapixant 50 mg BID on Days 1-3 and once daily in the morning Day 4 in Period 3
Period: Period 1
Arm/Group | Gefapixant 50 mg>Gefapixant 300 mg>Placebo | Gefapixant 50 mg>Placebo>Gefapixant 300 mg | Gefapixant 300 mg>Gefapixant 50 mg>Placebo | Gefapixant 300 mg>Placebo>Gefapixant 50 mg | Placebo> Gefapixant 50 mg>Gefapixant 300 mg | Placebo> Gefapixant 300 mg>Gefapixant 50 mg
Started | 3 | 4 | 3 | 3 | 3 | 4
Completed | 3 | 4 | 3 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Wash-out
Arm/Group | Gefapixant 50 mg>Gefapixant 300 mg>Placebo | Gefapixant 50 mg>Placebo>Gefapixant 300 mg | Gefapixant 300 mg>Gefapixant 50 mg>Placebo | Gefapixant 300 mg>Placebo>Gefapixant 50 mg | Placebo> Gefapixant 50 mg>Gefapixant 300 mg | Placebo> Gefapixant 300 mg>Gefapixant 50 mg
Started | 3 | 4 | 3 | 3 | 3 | 4
Completed | 3 | 4 | 3 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Gefapixant 50 mg>Gefapixant 300 mg>Placebo | Gefapixant 50 mg>Placebo>Gefapixant 300 mg | Gefapixant 300 mg>Gefapixant 50 mg>Placebo | Gefapixant 300 mg>Placebo>Gefapixant 50 mg | Placebo> Gefapixant 50 mg>Gefapixant 300 mg | Placebo> Gefapixant 300 mg>Gefapixant 50 mg
Started | 3 | 4 | 3 | 3 | 3 | 4
Completed | 3 | 4 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Period: Wash-out
Arm/Group | Gefapixant 50 mg>Gefapixant 300 mg>Placebo | Gefapixant 50 mg>Placebo>Gefapixant 300 mg | Gefapixant 300 mg>Gefapixant 50 mg>Placebo | Gefapixant 300 mg>Placebo>Gefapixant 50 mg | Placebo> Gefapixant 50 mg>Gefapixant 300 mg | Placebo> Gefapixant 300 mg>Gefapixant 50 mg
Started | 3 | 4 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Personal reasons | 0 | 1 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Gefapixant 50 mg>Gefapixant 300 mg>Placebo | Gefapixant 50 mg>Placebo>Gefapixant 300 mg | Gefapixant 300 mg>Gefapixant 50 mg>Placebo | Gefapixant 300 mg>Placebo>Gefapixant 50 mg | Placebo> Gefapixant 50 mg>Gefapixant 300 mg | Placebo> Gefapixant 300 mg>Gefapixant 50 mg
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gefapixant 50 mg>Gefapixant 300 mg>Placebo | Gefapixant 50 mg>Placebo>Gefapixant 300 mg | Gefapixant 300 mg>Gefapixant 50 mg>Placebo | Gefapixant 300 mg>Placebo>Gefapixant 50 mg | Placebo> Gefapixant 50 mg>Gefapixant 300 mg | Placebo> Gefapixant 300 mg>Gefapixant 50 mg | Total
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 4 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.7 (7.0) | 27.5 (7.6) | 43.3 (7.6) | 31.3 (8.0) | 52.7 (8.1) | 40.0 (14.3) | 38.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 0 | 1 | 2 | 7
  Male | 2 | 3 | 1 | 3 | 2 | 2 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 3 | 3 | 3 | 4 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 4 | 3 | 3 | 3 | 4 | 20
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Provocative Concentration (PC20) After Methacholine Challenge
Description: The provocative concentration (PC) of inhaled methacholine required to reduce forced expiratory volume in 1 second (FEV1) by 20% (PC20) was calculated from the methacholine challenge at screening and 2 hours (+15 minutes) post dose on Day 3 of each Treatment Period using a five-breath dosimeter method. The primary endpoint was the methacholine PC20 value normalized by means of a log (base 2) transformation, at 2 dose levels compared with placebo in participants with asthma following provocation with methacholine.
Time Frame: Screening (Day -21 to Day -1) and Day 3
Population: Analysis population included all randomized participants who received at least 1 dose of study medication and had any post-dose efficacy evaluations for a given Treatment Period and who completed all 3 Treatment Periods.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: log [mg/mL]
Groups:
- Gefapixant 50: Participants received gefapixant 50 mg twice daily for 3.5 days during one period of the study
- Gefapixant 300: Participants received gefapixant 300 mg twice daily for 3.5 days during one period of the study
- Placebo: Participants received placebo twice daily for 3.5 days during each period of the study
Arm/Group | Gefapixant 50 | Gefapixant 300 | Placebo
Number analyzed (Participants) | 18 | 18 | 18
log [mg/mL] | 0.91 (214.4) | 0.84 (181.0) | 0.82 (260.1)
Statistical Analysis 1: Comparison: Gefapixant 50 vs Placebo; Test type: Superiority; p = 0.616, ANOVA; Geometric means ratio = 1.108, 95% CI 2-sided [0.734 to 1.673] — Analysis was based on an ANOVA model with log (base 2) PC20 methacholine challenge at each period as dependent variable, treatment and period as fixed effects and participant as random effect
Statistical Analysis 2: Comparison: Gefapixant 300 vs Placebo; Test type: Superiority; p = 0.939, ANOVA; Geometric means ratio = 1.016, 95% CI 2-sided [0.673 to 1.534] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Gefapixant 50 vs Gefapixant 300; Test type: Superiority; p = 0.671, ANOVA; Geometric means ratio = 0.917, 95% CI 2-sided [0.607 to 1.384] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Highest FEV1 After Methacholine Challenge
Description: Serial FEV1 was measured post inhalation of methacholine challenges for 90 minutes. The highest FEV1 at 5, 15, 30, 45, 60, and 90 minutes following methacholine challenge were evaluated for each subject. The minimum highest FEV1 was derived using the first three available measures that cover the first 30 minutes after the challenge.
Time Frame: Screening (Day -21 to Day -1) and Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- Screening: Screening (Day -21 to Day -1)
Arm/Group | Screening | Gefapixant 50 | Gefapixant 300 | Placebo
Number analyzed (Participants) | 18 | 18 | 18 | 18
Liters
  + 5 minutes | 2.44 (0.66) | 2.53 (0.70) | 2.43 (0.71) | 2.54 (0.75)
  +15 minutes | 2.69 (0.75) | 2.72 (0.80) | 2.67 (0.83) | 2.77 (0.84)
  +30 minutes | 2.86 (0.82) | 2.93 (0.88) | 2.83 (0.86) | 2.94 (0.89)
  +45 minutes | 2.93 (0.83) | 3.02 (0.88) | 2.99 (0.90) | 3.03 (0.93)
  +60 minutes | 2.99 (0.84) | 3.11 (0.93) | 3.06 (0.91) | 3.14 (0.96)
  +90 minutes | 3.10 (0.88) | 3.15 (0.93) | 3.12 (0.90) | 3.18 (0.95)
  Minimum Highest FEV1 | 2.44 (0.66) | 2.53 (0.70) | 2.43 (0.71) | 2.54 (0.75)
Statistical Analysis 1: Comparison: Gefapixant 300 vs Placebo; Test type: Superiority; p = 0.066, ANOVA; Mean Difference (Final Values) = -0.111, 95% CI 2-sided [-0.230 to 0.008] — Analysis is based on an ANOVA model with minimum highest FEV1 after methacholine challenge at each period as dependent variable, treatment and period as fixed effects and participant as random effect
Statistical Analysis 2: Comparison: Gefapixant 50 vs Placebo; Test type: Superiority; p = 0.843, ANOVA; Mean Difference (Final Values) = -0.012, 95% CI 2-sided [-0.131 to 0.107] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Gefapixant 50 vs Gefapixant 300; Test type: Superiority; p = 0.098, ANOVA; Mean Difference (Final Values) = -0.099, 95% CI 2-sided [-0.218 to 0.020] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 42 days
Description: All cause mortality events were assessed for all randomized participants. Non-serious and Serious AEs were assessed for all participants who were randomized and received at least one dose of study drug.
Groups:
- Gefapixant 50 mg: Participants received gefapixant 50 mg twice daily for 3.5 days during one period of the study
- Gefapixant 300 mg: Participants received gefapixant 300 mg twice daily for 3.5 days during one period of the study
Arm/Group | Gefapixant 50 mg | Gefapixant 300 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 16/19 | 19/19 | 8/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefapixant 50 mg (N=19) | Gefapixant 300 mg (N=19) | Placebo (N=20)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Thirst (General disorders) | 1 (1) | 1 (1) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 13 (13) | 18 (18) | 0 (0)
Headache (Nervous system disorders) | 8 (9) | 6 (6) | 6 (6)
Hypogeusia (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No data collected as part of this study will be utilized in any written work, including publications, without the written consent of Sponsor.